CLINICAL TRIAL: NCT04916782
Title: Evaluation of Favorable Functional Recovery Predictors at 3 Months of Patients With Acute Ischemic Stroke Treated by Mechanical Thrombectomy
Brief Title: Evaluation of Functional Recovery of Patients With Acute Ischemic Stroke Treated by Thrombectomy
Acronym: EPIC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0393
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Acute Ischemic Stroke
Keywords: stroke; outcome; Thrombectomy
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group
  Interventions: Other: Quality of life Questionnaire

INTERVENTIONS:
Other: Quality of life Questionnaire — Quality of life questionnaire

SUMMARY:
The management of cerebral infarctions (CI) is a real public health issue. The French National Authority for Health recommends Mechanical Thrombectomy (MT) either in combination with Intravenous Thrombolysis (IVT), or alone, after failure of IVT or in case of contraindication to IVT, within 6 hours of the onset of symptoms.

The objective is to determine the factors predicting good functional recovery at 3 months in order to establish the typical profile of the "good responder" patient to MT and to evaluate functional recovery at 3 and 12 months (mRS ≤ 2) according to the modality of MT (depending on whether it is performed during the day or at night), the age of the patients, the equipment used for MT, the type of anaesthesia, as well as the impact of the metrics from the radiological evaluation in the patient's management. patient management.

DETAILED DESCRIPTION:
The management of cerebral infarction (CI) is a real public health issue. There are 120,000 hospitalizations of CI patients per year in France. It is the leading cause of acquired disability and the second leading cause of dementia. Since 2015, the scientific community has demonstrated the benefits of mechanical thrombectomy (MT) in the treatment of patients with CI. The French National Authority for Health (HAS) recommends MT either in combination with intravenous (IV) thrombolysis, or alone, after failure of IV thrombolysis or in case of contraindication to IV thrombolysis, within 6 hours of the onset of symptoms.

Based on previous studies, the HAS has extended its recommendations for the treatment of patients (with occlusion of large vessels of the anterior cerebral circulation) whose onset of symptoms or last seen asymptomatic is between 6 and 16 hours, and may even extend up to 24 hours depending on strict inclusion criteria.

These previous clinical trials have shown the remarkable efficacy of MT in CI patients under the age of 80. There are no clear recommendations for MT in patients over 80 years of age, and further research is needed to improve the safety of MT.

Further research is needed to improve patient selection in the elderly. Today, predictive factors impacting on functional recovery such as age, blood glucose, and NIHSS neurological severity score have been evaluated. However, no association between these factors during the course of treatment has been established to determine the clinical and radiological characteristics that define the standard profile of "good responders" to MT.

The cohort is a continuation of the data previously collected in a database of the Commission Nationale de l'Informatique et des Libertés (CNIL). This database reports a complete follow-up (clinical, imaging and MT procedure data) of patients, from admission to 3 months after their hospitalisation. Some results have already been published.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Indication for treatment with Mechanical Thrombectomy
* Imaging on admission (Scanner and/or Magnetic Resonance Imaging (MRI)) showing occlusion of a large intracranial artery intracranial artery (anterior, middle, posterior cerebral artery, basilar artery, vertebral vertebral artery)
* Health insurance coverage
* Obtaining the patient's consent

Exclusion Criteria:

* Patient with a serious intercurrent pathology impacting the vital prognosis in the short term and making it impossible to follow up at 3 months.
* Patients for whom follow-up will be impossible (foreign tourists)
* Patients of legal age (under guardianship, under curatorship, deprived of liberty)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with cerebral infarction treated in the acute phase by thrombectomy
Sampling Method: Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Determine the predictive factors of good functional recovery (modified Rankin Score (mRS) ≤ 2) at 3 months in order to establish the typical profile of the patient "good responder" to Mechanical Thrombectomy (MT) | At 3 months

SECONDARY OUTCOMES:
Evaluate functional recovery at 3 months (mRS ≤ 2) according to the modality of MT (depending on whether it is carried out during the day or at night) | At 3 months
Evaluate functional recovery at 12 months (mRS ≤ 2) according to the modality of MT (depending on whether it is carried out during the day or at night) | At 12 months
Evaluate functional recovery at 12 months (mRS ≤ 2) according to the age of the patients, specifically for the very elderly (> 80 years old) | At 12 months
Evaluate functional recovery at 3 months (mRS ≤ 2) according to the age of the patients, specifically for the very elderly (> 80 years old) | At 3 months
Evaluate functional recovery at 3 months (mRS ≤ 2) according to material used for MT | At 3 months
Evaluate functional recovery at 12 months (mRS ≤ 2) according to material used for MT | At 12 months
Evaluate functional recovery at 12 months (mRS ≤ 2) according to the type of anesthesia (conscious sedation / general anesthesia) | At 12 months
Evaluate functional recovery at 3 months (mRS ≤ 2) according to the type of anesthesia (conscious sedation / general anesthesia) | At 3 months
Evaluate functional recovery at 3 months (mRS ≤ 2) according to the impact of metrics from the radiological assessment in patient care | At 3 months
Evaluate functional recovery at 12 months (mRS ≤ 2) according to the impact of metrics from the radiological assessment in patient care | At 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France